CLINICAL TRIAL: NCT01550601
Title: Impact of the Preservation of the Gastric Antrum in the Technique of Sleeve Gastrectomy for the Treatment of the Morbid Obesity: a Prospective,Controlled, Randomized, Multicentrique Study.
Brief Title: Impact of the Preservation of the Gastric Antrum in the Technique of Sleeve Gastrectomy for the Treatment of the Morbid Obesity
Acronym: QUALISLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Marseille (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8643; 2010-A01021-38 (Other: ID-RCB)
Record Dates: First submitted 2012-02-27; First posted 2012-03-12 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Obesity, Morbid
Keywords: morbid obesity; gastrectomy; gastrinaemia; comorbidity; gastric antrum
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- bariatric surgery 1 (Other): Longitudinal gastrectomy (sleeve gastrectomy) is a technique of bariatric surgery. In this arm, patients have a bariatric surgery with conservation of gastric antrum.
  Interventions: Procedure: bariatric surgery
- bariatric surgery 2 (Experimental): Longitudinal gastrectomy (sleeve gastrectomy) is a technique of bariatric surgery. In this arm, patients have a bariatric surgery with ablation of gastric antrum.
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — The longitudinal gastrectomy (sleeve gastrectomy) is a technique of bariatric surgery recently validated (HAS on 2008).It consists of the realization of a partial gastrectomy of 2/3 (Fundus, gastric Body +/- antrum). However, lot of technical disagreements are brought back by expert teams. The most important disagreement concerns the conservation or the exeresis of the gastric antrum. In fact, the conservation of gastric antrum could facilitate the gastric emptying and to decrease the RGO (main complication) and act on the regulations of hormones modulators of the insulino-secretion.

SUMMARY:
The bariatric surgery is recognized, at present, as the only effective therapeutic for the patients with morbid obesity. Two surgical procedures (said restrictive) are considered as consensual: the adjustable calibrated horizontal gastroplasty under laparoscopy (ring périgastric) and Gastric Bypass under laparoscopy (LGBP). The longitudinal gastrectomy (sleeve gastrectomy) is a technique of bariatric surgery recently validated (HAS on 2008). It consists of the realization of a partial gastrectomy of 2/3 (Fundus, gastric Body +/- antrum). However, lot of technical disagreements are brought back by expert teams. The most important disagreement concerns the conservation or the exeresis of the gastric antrum. In fact, the conservation of gastric antrum could facilitate the gastric emptying and to decrease the RGO (main complication) and act on the regulations of hormones modulators of the insulino-secretion.

A prospective,randomized study comparing these both techniques is necessary to determine a unique consensual technique

DETAILED DESCRIPTION:
The main objective of this study is to compare the frequency of post-operative gastronomic appearance of gastroesophageal reflux(RGO) between two techniques of longitudinal gastrectomy under laparoscopy (gastrectomy coupling sleeve with antrum conservation or without antrum conservation) at patients with morbid obesity.

There are lot of secondary outcomes assessed in this study. In fact, one of secondary objectives is to compare between both techniques of longitudinal gastrectomy under laparoscopy described in the literature the efficiency on the loss of weight and global post-operative morbidity.

This study assess the impact of these surgery techniques on the comorbidity of the obesity and their treatments (type 2 diabetes, arterial hypertension, sleep apnea syndrome, arthralgia, dyslipemia).

ELIGIBILITY:
Inclusion Criteria:

Patients with an indication of bariatric surgery (Recommendations HAS) defined as follows:

* IMC = 40kg/m² with failure of the dietary treatments during at least 1 year, or
* IMC = 35kg/m ² if associated comorbidity (HTA, diabetes, gonarthrose, sleep apnea, dyslipidemia, severe respiratory diseases)
* Patients motivated by this surgery and to accept the post-operative constraints.
* Age: > 18 years and < 65 years.
* patient having received an favorable opinion to the multidisciplinary meeting
* patient with his/her consent.
* patient with French insurance

Exclusion Criteria:

* Women Patients presenting a current pregnancy (not effective contraception during the first year after surgery) or in age to procreate and without means of effective contraception (oestroprogestational)
* patient with a contraindication to the anesthesia
* patient with grave psychiatric disorders (psychotic, paranoid)
* Emotionally unstable Patient or showing psychiatric characteristics which according to the opinion of the psychologist or the surgeon are incompatible with this type of surgery
* patient with surgical histories esogastric
* Patient with an inflammation of the digestive system (severe esophagitis, gastrointestinal ulcer, CROHN disease)
* Patient with a severe cardiopulmonary affection or other severe organic affection
* patient with a risk of bleedings in the superior gastrointestinal part (esophageal varice)
* Patient with gastrointestinal congenital defects (stenosis, atresia)
* Patient with chronic alcoholism or drug addiction
* patient having a serious infection (HIV)
* Patient who refuses categorically the diet imposed by this surgery
* patient with a food of type "sweet eaters" (sweet food, high calorie liquid).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Comparison of the frequency appearance of RGO after surgery intervention (between two techniques longitudinal gastrectomy) in patients of morbid obesity | 12 months
  The main objective of this study is to compare the frequency of post-operative gastronomic appearance of gastroesophagal reflux(RGO) between both techniques of longitudinal gastrectomy under laparoscopy (gastrectomy coupling sleeve with antrum conservation or without antrum conservation) at patients with morbid obesity.

SECONDARY OUTCOMES:
Assessment of efficiency on loss of weight and global post-operative morbidity between both surgery techniques. | 12 months
  Comparison between both techniques of longitudinal gastrectomy under laparoscopy described in the literature in terms of efficiency on the loss of weight and global post-operative morbidity
Impact assessment of both types' surgery on the comorbidity and treatments of obesity | 12 months
  Assess the impact of these surgery techniques on the comorbidity of the obesity and their treatments (type 2 diabetes, arterial hypertension, sleep apnea syndrom, arthralgia, dyslipemia)
Assessment of gastrinemia between both groups (efficacy assessment) | at 1,3,12 months
  Assess the variations of the gastrinaemia according to the used technique (in fact, this hormone is partially secreted by the gastric antrum)

CONTACTS AND LOCATIONS:
Overall Officials: Nocca David, PU-PH, Principal Investigator — CHRU de Montpellier
Locations (1):
- CHRU Montpellier, Hopital Saint-Eloi, Montpellier, France